CLINICAL TRIAL: NCT03306602
Title: Clinical Evaluation of Bulk-fill vs Layered Composite Resin in Class I and II Posterior Restorations: A Randomized Controlled Pilot Study
Brief Title: Clinical Evaluation of Bulk-fill vs Layered Composite Resin in Class I and II Posterior Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Asst. Prof. Dr. NASIL SAKKIR, Assistant Professor, Department of Conservative Dentistry and Endodontics, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMMC/FOD/AR/B5/ E C-2017(26)
Record Dates: First submitted 2017-10-03; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Dental Caries Class I (Disorder); Dental Caries Class II
Keywords: Composite Resins; Dental Restorations

STUDY DESIGN:
Intervention Model Description: All the participants will receive both the experimental and control restoration. In the experimental cavity, Filtek Bulk Fill Posterior Restorative (3M ESPE) will be placed in 5 mm increments, eliminating the need for additional layers or multiple steps. The control restoration will be filled with Filtek Z350 XT (3M ESPE) using the 2 mm incremental layering technique.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The cavity in an individual will be randomly assigned to either the experimental or the control restoration, according to a predetermined scheme of randomization. If the participants have two cavities, they will not know in which cavity the experimental and control restoration were placed. All the restorations will be analyzed by using Modified United States Public Health Services (USPHS) criteria. The investigators and outcome assessors evaluating the restorations will not know which tooth has been restored with the experimental or control restoration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bulk Fill Composite (Experimental): In the experimental cavity, Filtek Bulk Fill Posterior Restorative (3M ESPE) will be placed in 5 mm increments, eliminating the need for additional layers or multiple steps.
  Interventions: Device: Filtek Bulk Fill Posterior Restorative
- Layered Composite (Active Comparator): The control restoration will be filled with Filtek Z350 XT (3M ESPE) using the 2 mm incremental layering technique.
  Interventions: Device: Filtek Z350 XT

INTERVENTIONS:
Device: Filtek Bulk Fill Posterior Restorative — Filtek™ Bulk Fill Posterior Restorative is a one-step bulk placement solution for fast and easy posterior resin restorations.
  Arms: Bulk Fill Composite
Device: Filtek Z350 XT — Filtek Z350XT is a material for incremental layered composite resin restorations
  Arms: Layered Composite

SUMMARY:
The aim of this study is to evaluate the clinical performance of Filtek Bulk Fill Posterior Restorative in Class I and Class II restorations compared to the conventional incremental technique using Filtek Z350XT over the period of 2 years. The null hypothesis of this study is that the bulk-fill composite will exhibit same result and clinical performance as conventional composite using incremental technique which has been used widely by dentists nowadays.

DETAILED DESCRIPTION:
In recent years, people are more concerned with the aesthetic qualities of dental restorations and in response to enhancements in the resin technologies, tooth-colored resin composite materials are increasingly being used for posterior teeth instead of amalgam fillings. Developments during the years in chemical composition, filler reinforcement, and adhesive techniques have resulted in many new modified categories of materials. Some researchers recommend the use of the incremental technique, in which the composite material is gradually placed in layers of 2mm or less.

This approach to restore teeth has a number of advantages, for example, it results in better light penetration and better polymerization of composite resin, reduction in cavity configuration factor, reduction in polymerization shrinkage stress and ensures that the resin adheres to the cavity walls. During curing of the resin, a network of polymers is formed, which becomes rigid due to increased cross linking of the polymer chains. Decreasing mobility of the network causes further shrinkage and results in a strain on the resin composite and cavity margins. The resulting stress has been associated with marginal deficiencies, enamel fractures, cuspal movement, and cracked cusps, which in turn may result in microleakage, post-operative sensitivity, and secondary caries. It has been stated that posterior class II and especially class I cavities with a high C-factor will result in greater stresses due to a larger number of bonded surfaces.

However, there are number of disadvantages associated with the use of an incremental approach to place the resin. For example, voids can be trapped in between the increments, bonding failure can occur in between the increments, difficulty in placing the composite material after cavity preparation and the long time taken for the procedure. In an effort to counter these problems, a new restorative material has been introduced in 2009 which is known as 'bulk-fill' composite, in order to increase efficiency of the operator. However, many clinicians who have accustomed to the incremental cure philosophy when placing the light-cured composite quite rightly question what has been changed to make these bulk-fill light-cured composite a variable alternative. According to some researchers, bulk-fill composite offers more advantages compared to the layered composite. These include increased efficiency in working time, reduced polymerization shrinkage and reduces the risk of contamination and voids forming between the resins.

The aim of this study is to evaluate the clinical performance of bulk-fill composite as compared to the layered composite technique in class I and class II restorations over the period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

Patient presenting with:

1. Any permanent premolar and molar requiring class I or II restorations;
2. Good oral hygiene;
3. Teeth in occlusion having at least one proximal contact with adjacent tooth;
4. Absence of any periodontal or pulpal pathology;
5. Absence of pain from the tooth to be restored;
6. Possible application of rubber dam during treatment

Exclusion Criteria:

1. Participants with unerupted tooth or partially erupted tooth,
2. Smoking,
3. Pregnant patients,
4. Severe bruxism habit,
5. Pathological pulpal or periodontal problems,
6. Fractured or visibly cracked teeth.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
Modified United States Public Health Services (USPHS) criteria | 2 years
  All the restorations will be analyzed by using Modified United States Public Health Services (USPHS) criteria, focusing more on the clinical criteria of the restoration. The characteristics of all the restorations will be described by using descriptive statistics using cumulative frequency distributions of the scores.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Abdul Rashid Hj Ismail, BDS,MSc,DDPH, Study Chair — Melaka Manipal Medical College
Locations (1):
- Melaka Manipal Medical College, Melaka Tengah, Melaka, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Dijken JW, Pallesen U. Randomized 3-year clinical evaluation of Class I and II posterior resin restorations placed with a bulk-fill resin composite and a one-step self-etching adhesive. J Adhes Dent. 2015 Feb;17(1):81-8. doi: 10.3290/j.jad.a33502. PMID 25625133
- [Background] van Dijken JW, Pallesen U. Posterior bulk-filled resin composite restorations: A 5-year randomized controlled clinical study. J Dent. 2016 Aug;51:29-35. doi: 10.1016/j.jdent.2016.05.008. Epub 2016 May 26. PMID 27238052
- [Background] van Dijken JW, Pallesen U. A randomized controlled three year evaluation of "bulk-filled" posterior resin restorations based on stress decreasing resin technology. Dent Mater. 2014 Sep;30(9):e245-51. doi: 10.1016/j.dental.2014.05.028. Epub 2014 Jun 21. PMID 24958689
- See also: Modified United States Public Health Service (USPHS) Ryge Criteria for Direct Clinical Evaluation of Restoration — http://multimedia.3m.com/mws/media/295038O/ryge-criteria-for-direct-clinical-evaluation-of-restoration.pdf?&fn=usphs_ryge_criteria.pdf.